CLINICAL TRIAL: NCT06342453
Title: CREATE: Clinical Research Examining the Arts as Targeted Elements in Childhood Cancer Care
Brief Title: CREATE: Art for Children With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jenny Raybin, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00026814; R34AT012497 (NIH); NCI-2024-01534 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00026814 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-03-05; First posted 2024-04-02 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Art Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I (focus group) (Active Comparator): Patients participate in focus groups to develop CrA intervention on study.
  Interventions: Procedure: Discussion; Other: Survey Administration
- Phase II arm I (CrA) (Experimental): Patients participate in CrA interventions comprising drawing, painting, and making sculptures with a trained artist for 30 minutes once a week for 4 sessions over 12 weeks.
  Interventions: Procedure: Art Therapy; Other: Survey Administration
- Phase II arm II (watch videos) (Active Comparator): Patients passively watch videos for 30 minutes once a week for 4 sessions over 12 weeks.
  Interventions: Other: Media Intervention; Other: Survey Administration

INTERVENTIONS:
Procedure: Art Therapy — Participate in CrA
  Arms: Phase II arm I (CrA)
Procedure: Discussion — Participate in art focus group, art-making
  Other Names: Discuss, creating art
  Arms: Phase I (focus group)
Other: Media Intervention — Watch videos
  Arms: Phase II arm II (watch videos)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial is being done to develop and test how well creative arts interventions (drawing, painting, making sculptures) compared to watching videos can affect symptoms and impact the quality of life in children with cancer. Creative arts mind-body interventions (CrA) are one type of complementary health interventions which have been associated with improved quality of life and reduced symptom burden among children with cancer. CrA is an ideal intervention for children with cancer due to the long hours spent in the hospital setting for treatments, the creativity and developmental focus of children, and their potential ability to communicate more easily through art than words. Researchers want to develop and test a CrA intervention to help improve symptoms and the quality of life of children with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Feasibility of an randomized controlled trial (RCT) of art among children with cancer.

SECONDARY OBJECTIVES:

I. Achieve recruitment rate target. II. Achieve accrual target. III. Achieve fidelity to intervention. IV. Assess initial effect sizes.

OUTLINE:

PHASE I: Patients participate in focus groups to develop CrA intervention on study.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients participate in CrA interventions comprising drawing, painting, and making sculptures with a trained artist for 30 minutes once a week for 4 sessions over 12 weeks.

ARM II: Patients passively watch videos for 30 minutes once a week for 4 sessions over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7 to 14 years of age
* Have been diagnosed with cancer of any type in the prior 12 months
* Be English literate (we will amend this criterium when the study surveys are validated in Spanish). Parent/caregiver of child participant may be Spanish speaking
* Physically and cognitively able to participate in creative arts
* Expected to receive enough treatment at local site to participate in all four intervention sessions

Exclusion Criteria:

* Not English literate
* Otherwise unable to complete study procedures

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants that complete all interventions and data collection time points | Up to day 90
  Will be considered feasible if 80% of participants complete 4 intervention sessions and 3 data collection time points. Will be summarized across and within each study arm using means and standard deviations for continuous variables, and frequency counts and percentages for nominal variables.

SECONDARY OUTCOMES:
Number of eligible participants that enroll in the study (feasibility threshold of 80%) | Up to to 24 months
  Will use 95% confidence intervals to estimate the precision of all point estimates.
Number of participants that complete all interventions and all surveys in the study. | Up to 24 months
  Goal of 80% of recruited participants. Will use 95% confidence intervals to estimate the precision of all point estimates.
Number of intervenor fidelity surveys that obtain at least 95% score. | Up to 24 months
  Will use 95% confidence intervals to estimate the precision of all point estimates.
Comparison of scores on the PRO-CTCAE between intervention arms | Up to 24 months
  Will use National Cancer Institute's Pediatric Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). The PRO-CTCAE Measurement System characterizes the frequency, severity, interference, and presence/absence of symptomatic toxicities. Answers ranging from None to Very Severe (none=0 to very severe=4); Not at All to Very Much (not at all=0 to very much=4), Never to Almost Constantly (0=never to almost constantly=4). Will be assessed by comparing outcome measure results between arms. Will use 95% confidence intervals to estimate the precision of all point estimates.
Comparison of scores on the PROMIS between intervention arms | Up to 24 months
  Will use PROMIS Pediatric Global Health-7 measure, a brief 7-item summary assessment of a child's self-reported health. This measure contains 7 items assessing global health (physical and mental wellbeing. All items are completed on a 5-point Likert scale (1= Poor to 5 = Excellent, or 1 = Never to 5 = Always or Almost always, depending on the domain). Will be assessed by comparing outcome measure results between arms. Will use 95% confidence intervals to estimate the precision of all point estimates.
Comparison of scores on the Faces between intervention arms | Up to 24 months
  Will be assessed using a Faces scale with 9 faces in order of happy to sad to assess emotional reactions. Will be assessed by comparing outcome measure results between arms. Will use 95% confidence intervals to estimate the precision of all point estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Raybin, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share by publishing in an ICMJE journal and will also submit data and metadata to the Dyad data repository.